CLINICAL TRIAL: NCT03017261
Title: TSolution One® Total Knee Arthroplasty Clinical Trial
Brief Title: TSolution One® Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Think Surgical Inc. (Industry)
Collaborators: MCRA (Industry); Medical Metrics Diagnostics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-PROTO-01
Record Dates: First submitted 2016-12-19; First posted 2017-01-11 (Estimated); Results first posted 2020-05-22 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-05

CONDITIONS: Osteoarthritis, Knee
Keywords: Osteoarthritis; Arthroplasty; Robotic Surgery; Knee
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- TSolution One® (Experimental): This group will undergo total knee arthroplasty with the TSolution One® System for the preparation of the femoral and tibial cuts.
  Interventions: Device: TSolution One®

INTERVENTIONS:
Device: TSolution One® — Total knee arthroplasty with the TSolution One® System for the preparation of the femoral and tibial cuts.

SUMMARY:
The goal of this prospective, non-randomized, multicenter clinical trial is to determine whether robotic-assisted total knee arthroplasty performed with TSolution One® System is safe and effective for use as an alternative to the conventional manual techniques. Clinical and radiographic outcomes for robotic-assisted total knee arthroplasty performed with the TSolution One® System will be collected preoperatively, intraoperatively, and postoperatively up to a follow-up period of no less than 6 months and no more than 12 months. These outcomes will be compared to the ones reported in the literature for conventional manual techniques.

DETAILED DESCRIPTION:
This clinical investigation will be conducted as a prospective, non-randomized, multicenter study. The primary objective of this study is to demonstrate that the TSolution One System is safe and effective for use as an alternative to manual planning and sawing/cutting techniques. The primary effectiveness objective of this study is to demonstrate that the TSolution One® System is effective for use as an alternative to manual planning and sawing/cutting techniques by comparing the rate of malalignment for mechanical axis greater than 3° at 3 months to the rate reported in the literature (i.e. 32%) and to demonstrate significant clinical benefit by reducing the number of malaligned patients by at least 50% (i.e. from 32% to ≤ 16%). The safety objective of this study is based on the rate of intraoperative and postoperative TKA complications, with a follow-up period of no less than 6 months and no more than 12 months, and to compare this rate to the rate reported in the literature. The secondary objective of this study is to summarize the distribution of improvements in patients' self-reported assessment of postoperative function and quality-of-life from baseline to a maximum of 12 months. Additionally, other preoperative planning alignment goals (e.g. Knee V-V Alignment; Femoral Joint Line Alignment Angle; Tibial Joint Line Alignment Angle; Tibial Slope Angle) will be compared to the post-operative alignment at 3 months.

Investigators will recruit subjects from patients in their practice who require unilateral total knee arthroplasty. Patients will be screened to identify eligible candidates based on the inclusion and exclusion criteria. A total of one hundred fifteen (115) patients will be enrolled in the study across the participating sites. All patients will sign an informed consent form prior to participating in the study.

Prior to undergoing the investigational procedure, the patients will complete baseline surveys of function and quality of life (Knee Society Score survey and the SF-12 Health Survey) and have baseline radiographs and a CT scan of the knee.

Each patient will then undergo robotic-assisted total knee arthroplasty with the TSolution One® System. The investigators will evaluate intra- and postoperative complications. Postoperative radiographs and a CT scan will be used to measure limb alignment using a standardized radiographic evaluation protocol. Each patient will complete a postoperative Knee Society Score survey and the SF-12 Health Survey to assess functional outcomes and quality-of-life following the investigational procedure.

ELIGIBILITY:
Inclusion Criteria:

1. At least 21 years of age.
2. Skeletally mature, as evidenced by closed epiphyses.
3. Eligible for primary unilateral TKA due to osteoarthritis defined radiographically by a Kellgren-Lawrence Grade of 3 or higher.
4. Able to understand and willing to comply with the requirements of the study.
5. Able to give voluntary, written informed consent to participate and has signed an Informed Consent Form specific to this study.

Exclusion Criteria:

1. Has undergone previous open knee surgery in the operative knee.
2. Has a body mass index (BMI) > 40 kg/m2.
3. Is a candidate for bilateral TKA.
4. Has a coronal deformity greater than 20° or a sagittal flexion contracture greater than 15°.
5. Has an active systemic infection or an active local infection in or near the operative knee joint, or has a previous history of joint infection.
6. Has a pathological skeletal condition or skeletal immaturity which would significantly compromise the ability of the bone to withstand the stress required for preparation of the bones and proper implantation of the prostheses (e.g., severe osteoporosis, Paget's disease, renal osteodystrophy, AVN, sickle cell disease, etc.).
7. Has femoral or tibial bone stock that is of poor quality or inadequate to provide stability for femoral or tibial fixation.
8. Has any type of metallic implant in the operative leg.
9. Has a known or suspected sensitivity to any of the materials in the investigational device or implant components (i.e. cobalt, chromium, titanium, stainless steel, titanium nitride, aluminum, polyethylene, PVC plastic)
10. Has a systemic illness or a neuromuscular, neurosensory, or musculoskeletal deficiency that would render the patient unable to perform appropriate postoperative rehabilitation.
11. Has a neuromuscular disorder that would create an unacceptable risk of prosthesis instability or fixation failure.
12. Has significant comorbidities or conditions associated with high risk for surgical or anesthetic survival (e.g. peripheral vascular disease, unstable cardiac disease, poorly controlled diabetes, immunosuppression, etc.).
13. Is pregnant or intends to become pregnant during the course of the study.
14. Has previously experienced a stroke.
15. Is participating concurrently in another clinical trial, or has participated in a clinical trial within the last 90 days, or intends to during the course of the study.
16. Has a medical or psychiatric condition which, in the opinion of the investigator, poses a risk of the patient being unable to complete the study or presents risks associated with study participation.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2017-02-18 (Actual); Primary Completion 2019-06-26 (Actual); Study Completion 2019-06-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bernard N Stulberg, MD, Principal Investigator — St. Vincent Charity Medical Center
Locations (6):
- United States (6):
  - Hackensack University Medical Center, Hackensack, New Jersey
  - NYU Langone Medical Center, New York, New York
  - St. Francis Hospital, The Heart Center®, Roslyn, New York
  - North Carolina Specialty Hospital, Durham, North Carolina
  - St. Vincent Charity Medical Center, Cleveland, Ohio
  - Houston Methodist West Hospital, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: 6 Week Follow up
Arm/Group | TSolution One®
Started | 115
Completed (8 did not complete the procedure with the device leaving 107 in the per protocol cohort.) | 115
Not Completed | 0
Period: 3 Month Follow up
Arm/Group | TSolution One®
Started | 115
Completed | 115 (1 failed to compete 3M imaging so only 114 have 3M data for tibial slope and KSS Objective Score.)
Not Completed | 0
Period: 6 Month Follow up
Arm/Group | TSolution One®
Started | 115
Completed (2 failed to compete 6M imaging so only 104 have 6M data for KSS Objective Score.) | 106
Not Completed | 9
Period: 12 Month Follow up
Arm/Group | TSolution One®
Started | 106
Completed | 59 (1 failed to compete 12M imaging so only 58 have 12M data for KSS Objective Score.)
Not Completed | 47

BASELINE CHARACTERISTICS:
Arm/Group | TSolution One®
Number analyzed (Participants) | 115
Age, Continuous [Mean (Standard Deviation); unit: years] — Age at surgery
  years | 65.91 (8.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57
  Male | 58
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9
  Not Hispanic or Latino | 106
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 10
  White | 96
  More than one race | 0
  Unknown or Not Reported | 7
Region of Enrollment [Number; unit: participants]
  United States | 115

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Postoperative Coronal Limb Alignment More Than ±3 Deg From the Planned Coronal Limb Alignment
Description: Comparison between planned and postoperative coronal limb alignment assessed as the difference between the planned hip-knee-ankle angle and the achieved hip-knee-ankle angle after surgery.
Time Frame: 3 months follow-up
Population: 8 patients did not complete the surgical procedure with the investigational device and were not included in the per protocol cohort.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | TSolution One®
Number analyzed (Participants) | 107
percentage of patients | 11.2 [6.3 to 18.2]

2. Primary Outcome: Adverse Events
Description: Adverse events will be assessed as the percentage of patients with TCAT (TSolutionOne Computer Assisted Tool)-assisted implantation experiencing the composite safety endpoint of typical adverse events
Time Frame: Up to 12 months follow-up
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | TSolution One®
Number analyzed (Participants) | 107
Participants | 0

3. Secondary Outcome: Percentage of Patients Experiencing a Composite of Relevant Safety Adverse Events
Description: Adverse events assessed as the percentage of patients with TCAT (TSolutionOne Computer Assisted Tool)-assisted implantation experiencing the composite safety endpoint of typical adverse events.
Time Frame: Up to 12 months follow-up
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | TSolution One®
Number analyzed (Participants) | 107
Participants | 0

4. Secondary Outcome: Bleeding Complications
Description: Number of patients experiencing bleeding complications will be assessed based on the incidence of transfusions required (autologous or allogenic).
Time Frame: Up to 12 months follow-up
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | TSolution One®
Number analyzed (Participants) | 107
Participants | 0

5. Secondary Outcome: Change in (KSS) Knee Society Objective Score From Baseline
Description: The computed difference in the total KSS objective score measured before surgery and after the surgery at this timepoint. The minimum KSS objective score is 0. The typical maximum KSS objective score is approximately 105 and depends on patient anatomy. Lower scores indicate a less functional knee joint reported as the result of an examination performed by a surgeon. The outcome measure reported is the difference between the objective score measured prior to surgery and the objective score measured at this time point.
Time Frame: Baseline to 6 Weeks
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | TSolution One®
Number analyzed (Participants) | 115
Units on a scale | 39.1 (19.7)

6. Secondary Outcome: Change in Knee Society Objective Score From Baseline
Description: as for outcome 5
Time Frame: Baseline to 3 Months
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | TSolution One®
Number analyzed (Participants) | 114
Units on a scale | 44.1 (19.1)

7. Secondary Outcome: Change in Knee Society Objective Score From Baseline
Description: as for outcome 5
Time Frame: Baseline to 6 Months
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | TSolution One®
Number analyzed (Participants) | 104
Units on a scale | 46.4 (18)

8. Secondary Outcome: Change in Knee Society Objective Score From Baseline
Description: as for outcome 5
Time Frame: Baseline to 12 Months
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | TSolution One®
Number analyzed (Participants) | 58
Units on a scale | 48.2 (18)

9. Secondary Outcome: Change in Knee Society Satisfaction Score From Baseline
Description: The computed difference in the total KSS satisfaction score measured before surgery and after the surgery at this timepoint. The minimum KSS satisfaction score is 0. The maximum KSS satisfaction score is 40. Lower scores indicate lower levels of patient reported satisfaction with knee pain and function. The outcome measure reported is the difference between the satisfaction score measured prior to surgery and the satisfaction score measured at this time point.
Time Frame: Baseline to 6 Weeks
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | TSolution One®
Number analyzed (Participants) | 115
Units on a scale | 12.3 (10.3)

10. Secondary Outcome: Change in Knee Society Satisfaction Score From Baseline
Description: as for outcome 9
Time Frame: Baseline to 3 Months
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | TSolution One®
Number analyzed (Participants) | 115
Units on a scale | 16.2 (10.2)

11. Secondary Outcome: Change in Knee Society Satisfaction Score From Baseline
Description: as for outcome 9
Time Frame: Baseline to 6 Months
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | TSolution One®
Number analyzed (Participants) | 106
Units on a scale | 18.1 (9.2)

12. Secondary Outcome: Change in Knee Society Satisfaction Score From Baseline
Description: as for outcome 9
Time Frame: Baseline to 12 Months
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | TSolution One®
Number analyzed (Participants) | 59
Units on a scale | 20.2 (9.5)

13. Secondary Outcome: Change in Knee Society Functional Score From Baseline
Description: The computed difference in the total KSS functional score measured before surgery and after the surgery at this timepoint. The minimum KSS functional score is 0. The maximum KSS satisfaction score is 100. Lower scores indicate increased functional limitations reported by patients. The outcome measure reported is the difference between the functional score measured prior to surgery and the functional score measured at this time point.
Time Frame: Baseline to 6 Weeks
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | TSolution One®
Number analyzed (Participants) | 115
Units on a scale | 13.2 (20.3)

14. Secondary Outcome: Change in Knee Society Functional Score From Baseline
Description: as for outcome 13
Time Frame: Baseline to 3 Months
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | TSolution One®
Number analyzed (Participants) | 115
Units on a scale | 25.2 (21.3)

15. Secondary Outcome: Change in Knee Society Functional Score From Baseline
Description: as for outcome 13
Time Frame: Baseline to 6 Months
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | TSolution One®
Number analyzed (Participants) | 106
Units on a scale | 34.2 (19.6)

16. Secondary Outcome: Change in Knee Society Functional Score From Baseline
Description: as for outcome 13
Time Frame: Baseline to 12 Months
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | TSolution One®
Number analyzed (Participants) | 59
Units on a scale | 42.3 (18.1)

17. Secondary Outcome: Pre-operative (KSS) Knee Society Patient Expectation Score
Description: Patient reported expectations for anticipated improvement in pain level and increase in activities as a result of planned knee replacement surgery. Expectations are reported on a scale of 0-15 where higher numbers indicate higher patent expectations. A score of 0 indicates that a patient had no expectations. A score of 15 indicates the highest level of expectations.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | TSolution One®
Number analyzed (Participants) | 115
Units on a scale | 14.5 (1)

18. Secondary Outcome: Post-operative (KSS) Knee Society Patient Expectation Score
Description: Patient reported evaluation of improvement in pain level and increase in activities after knee replacement surgery as compared to their pre-operative expectations. Expectations are reported on a scale of 0-15 where higher numbers indicate more fully met or exceeded expectations. A score of 0 indicates that none of the patient's pre-operative expectations were met. A score of 15 indicates that all of the patient's pre-operative expectations were exceeded.
Time Frame: 6 Weeks
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | TSolution One®
Number analyzed (Participants) | 115
Units on a scale | 9.8 (3.2)

19. Secondary Outcome: Post-operative (KSS) Knee Society Patient Expectation Score
Description: as for outcome 18
Time Frame: 3 Months
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | TSolution One®
Number analyzed (Participants) | 115
Units on a scale | 10.1 (3.0)

20. Secondary Outcome: Post-operative (KSS) Knee Society Patient Expectation Score
Description: as for outcome 18
Time Frame: 6 Months
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | TSolution One®
Number analyzed (Participants) | 106
Units on a scale | 10.3 (3.1)

21. Secondary Outcome: Post-operative (KSS) Knee Society Patient Expectation Score
Description: as for outcome 18
Time Frame: 12 Months
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | TSolution One®
Number analyzed (Participants) | 59
Units on a scale | 11.3 (2.7)

22. Secondary Outcome: Change in SF-12 (Short-form 12 Question) Physical Component Score From Baseline
Description: The computed difference in the total SF-12 physical component score measured before surgery and after the surgery at this timepoint. The minimum SF-12 physical component score is 0. The maximum SF-12 physical component score is 100. Lower scores indicate lower levels of patient reported physical health reported by patients The outcome measure reported is the difference between the SF-12 physical component score measured prior to surgery and the SF-12 physical component score measured at this time point.
Time Frame: Baseline to 6 Weeks
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | TSolution One®
Number analyzed (Participants) | 115
Units on a scale | 4.6 (11.2)

23. Secondary Outcome: Change in SF-12 (Short-form 12 Question) Physical Component Score From Baseline
Description: as for outcome 22
Time Frame: Baseline to 3 Months
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | TSolution One®
Number analyzed (Participants) | 115
Units on a scale | 10.6 (10.4)

24. Secondary Outcome: Change in SF-12 (Short-form 12 Question) Physical Component Score From Baseline
Description: as for outcome 22
Time Frame: Baseline to 6 Months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | TSolution One®
Number analyzed (Participants) | 106
Units on a scale | 13.3 (11.4)

25. Secondary Outcome: Change in SF-12 (Short-form 12 Question) Physical Component Score From Baseline
Description: as for outcome 22
Time Frame: Baseline to 12 Months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | TSolution One®
Number analyzed (Participants) | 59
Units on a scale | 15.9 (10.5)

26. Secondary Outcome: Change in SF-12 (Short Form 12 Question) Mental Component Score From Baseline
Description: The computed difference in the total SF-12 physical component score measured before surgery and after the surgery at this timepoint. The minimum SF-12 physical component score is 0. The maximum SF-12 physical component score is 100. Lower scores indicate lower levels of patient reported mental health reported by patients The outcome measure reported is the difference between the SF-12 physical component score measured prior to surgery and the SF-12 physical component score measured at this time point.
Time Frame: Baseline to 6 Weeks
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | TSolution One®
Number analyzed (Participants) | 115
Units on a scale | -2.0 (10.9)

27. Secondary Outcome: Change in SF-12 (Short-form 12 Question) Mental Component Score From Baseline
Description: as for outcome 26
Time Frame: Baseline to 3 Months
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | TSolution One®
Number analyzed (Participants) | 115
Units on a scale | 0.4 (10.5)

28. Secondary Outcome: Change in SF-12 (Short-form 12 Question) Mental Component Score From Baseline
Description: as for outcome 26
Time Frame: Baseline to 6 Months
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | TSolution One®
Number analyzed (Participants) | 106
Units on a scale | 1.4 (9.6)

29. Secondary Outcome: Change in SF-12 (Short-form 12 Question) Mental Component Score From Baseline
Description: as for outcome 26
Time Frame: Baseline to 12 Months
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | TSolution One®
Number analyzed (Participants) | 59
Units on a scale | 2.9 (11.0)

30. Secondary Outcome: Tibial Joint Line Alignment Angle (TJLA) Change From Pre-op Plan
Description: Comparison between planned and postoperative TJLA will be assessed as the difference between the planned TJLA angle and the achieved TJLA angle after surgery.
Time Frame: Baseline to 3 Months
Measure: Mean (Standard Deviation); unit: Angle
Arm/Group | TSolution One®
Number analyzed (Participants) | 115
Angle | .35 (1.64)

31. Secondary Outcome: Femoral Joint Line Alignment Angle (FJLA) Change From Pre-op Plan
Description: Comparison between planned and postoperative FJLA will be assessed as the difference between the planned FJLA angle and the achieved FJLA angle after surgery.
Time Frame: Baseline to 3 Months
Measure: Mean (Standard Deviation); unit: Angle
Arm/Group | TSolution One®
Number analyzed (Participants) | 115
Angle | -0.93 (1.29)

32. Secondary Outcome: Tibial Slope Change From Pre-op Plan
Description: Comparison between planned and postoperative Tibial Slope will be assessed as the difference between the planned Tibial Slope and the achieved Tibial Slope after surgery.
Time Frame: Baseline to 3 Months
Measure: Mean (Standard Deviation); unit: Angle
Arm/Group | TSolution One®
Number analyzed (Participants) | 114
Angle | -0.01 (1.53)

ADVERSE EVENTS:
Time Frame: 6 months for all subjects. 12 Months for those subjects that completed 12 months of follow-up.
Description: AE: Untoward medical occurrence, disease, injury, or untoward clinical signs, whether related or unrelated to the investigational device or its use.
  SAE: AE which: Led to a death, Resulted in: life threatening illness or injury, patient hospitalization or prolongation of existing hospitalization, patient disability or permanent damage or required intervention to prevent permanent impairment/damage, Led to a congenital abnormality or birth defect
Arm/Group | TSolution One®
All-Cause Mortality (participants affected / at risk) | 0/115
Serious Adverse Events (participants affected / at risk) | 12/115
Other Adverse Events (participants affected / at risk) | 55/115
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TSolution One® (N=115)
Stiffness of the joint (Musculoskeletal and connective tissue disorders) | 3 (3) — Index Side
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) — Non-index side
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Congestive Heart Failure (Cardiac disorders) | 1 (1)
Non-malignant asbestosis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hip Fracture (Musculoskeletal and connective tissue disorders) | 1 (1) — Due to injury
Finger Fracture (Musculoskeletal and connective tissue disorders) | 1 (1) — Due to injury
Phimosis (Renal and urinary disorders) | 1 (1) — With difficulty urinating
Proctocolitis (Gastrointestinal disorders) | 1 (1) — with diverticulitis
Gastrointestinal Bleed (Gastrointestinal disorders) | 1 (1)
Dehydration (General disorders) | 1 (1)
Breast Cancer (Reproductive system and breast disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TSolution One® (N=115)
Anal Fissure (Skin and subcutaneous tissue disorders) | 1 (1)
Arrhythmia (Cardiac disorders) | 2 (2)
Back Pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) — With neck pain
Bladder Infection (Infections and infestations) | 1 (1)
Bleeding, unrelated to surgical site/procedure (Vascular disorders) | 1 (1) — Nose bleed
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) — With shortness of breath
Deep Vein Thrombosis (Vascular disorders) | 1 (1) — Index Side
Delayed Wound Healing (General disorders) | 2 (2)
Dental Infection (Infections and infestations) | 1 (1)
Dental Pain (General disorders) | 1 (1)
Difficulty Breathing (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Edema (General disorders) | 5 (5) — Index side
Edema (General disorders) | 1 (1) — Non-index side
Edema (General disorders) | 1 (1) — Lower Extremity
Effusion (General disorders) | 4 (5) — Index Side
Exacerbation of anemia (Blood and lymphatic system disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (2) — Due to prescribed narcotics
Fall (Injury, poisoning and procedural complications) | 4 (4) — Due to injury
Fatigue (General disorders) | 2 (2)
Generalized anxiety disorder (Psychiatric disorders) | 1 (1)
Hernia (Musculoskeletal and connective tissue disorders) | 1 (1)
Hip pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Index knee pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Index knee pain (Injury, poisoning and procedural complications) | 1 (1) — Due to injury
Insect bite (General disorders) | 1 (1)
Nasal polyps (General disorders) | 1 (1)
MCL Injury (Injury, poisoning and procedural complications) | 1 (1) — Due to injury
Lichen Sclerosis (Skin and subcutaneous tissue disorders) | 1 (1)
Kidney Stone (Psychiatric disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Non-index knee pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) — Index side
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 4 (4) — Non-index side
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) — Cervical
Otitis media (Ear and labyrinth disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) — Surgical site
Pressure sores (Skin and subcutaneous tissue disorders) | 1 (1) — Surgical site
Rheumatoid Arthritis (Immune system disorders) | 1 (1)
Retained device pins (Injury, poisoning and procedural complications) | 1 (1) — Surgical site
Respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 2 (2) — Upper
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Seroma (General disorders) | 1 (1) — Index side
Seroma (General disorders) | 1 (1) — Surgical site
Systemic Infection (Infections and infestations) | 2 (2)
Surgical Incision Infection (Infections and infestations) | 2 (2)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 2 (2)
Thigh pain (Musculoskeletal and connective tissue disorders) | 1 (1) — Index side
Temporary hearing loss (Ear and labyrinth disorders) | 1 (1)
Toe fungus (Infections and infestations) | 1 (1)
Umbilical hernia (Musculoskeletal and connective tissue disorders) | 1 (1)
Worsening of Parkinson's Disease (Nervous system disorders) | 1 (1)
Urinary tract infection (Renal and urinary disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Pain (other musculoskeletal) (Musculoskeletal and connective tissue disorders) | 1 (1) — Gout
Pain (other musculoskeletal) (Musculoskeletal and connective tissue disorders) | 1 (1) — Bruise due to injury

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI must submit proposed publications to Sponsor for review per contract timelines.

Hospital & PI shall:

* not publish the Hospital's and PI's results until a multi-center publication is released; however, if a multi-center publication is not released within 1 year after the study, Hospital & PI may publish the results of their activities.
* keep all unpublished data & results confidential and not disclose such in greater detail than disclosed in any publications, presentations or disclosures.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-09): https://cdn.clinicaltrials.gov/large-docs/61/NCT03017261/Prot_SAP_000.pdf